CLINICAL TRIAL: NCT04059432
Title: CHAIN1 : Dental Wear and Musculoskeletal Disorders - Association?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Mainjot Amélie, DDS, MSc, PhD, University of Liege
Other Study IDs: CH001
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Tooth Wear; Musculoskeletal Disorder
Keywords: Tooth Wear; Musculoskeletal Disorders
MeSH Terms: conditions — Tooth Wear; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tooth Wear and Musculoskeletal Disorders evaluation — Evaluation of dental wear by BEWE (Basic Erosive Wear Examination: score 0-3) examination and Musculoskeletal disorders are listed by the "NORDIC" questionnaire developed by Kuorinka et al. (2001)

SUMMARY:
This study aims to explore the relationships between tooth wear (TW) and musculoskeletal disorders (MSDs). The null hypothesis is that TW is not associated to MSDs. It also explores the influence of bruxism signs, life habits and stress on TW and MSDs.

DETAILED DESCRIPTION:
This study is based on questionnaires and clinical examination performed by a dentist.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years old
* Have the mental abilities to participate in study
* Understand the language of the survey (French)
* Sign free and informed consent

Exclusion Criteria:

* Consult for a painful dental emergency
* Do not have at least 8 teeth per maxilla, with natural dental tissues in contact with the antagonistic teeth
* Being in the process of an orthodontic treatment
* Wear of a bimaxillary orthognathic nightguard

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients consulting in the Fixed Prosthesis Department (Dentistry Department) at the Polyclinic Lucien Brull from Liège University Hospital between March 2019 and October 2019
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Presence of musculoskeletal disorders (MSDs) | through study completion, an average of 1 year
  "Nordique Questionnaire": validated self-report questionnaire to evaluate musculo skeletal health, particularly MSD on 9 different zones
Tooth wear following BEWE index | through study completion, an average of 1 year
  Clinical examination will give a global score on 18 following Basic Erosive Wear Examination (BEWE) index.

SECONDARY OUTCOMES:
Life habits and stress | through study completion, an average of 1 year
  10-points likert scale self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Mainjot, Study Director — CHU-ULg
Locations (1):
- Institute of Dentistry University of Liege, Liège, Choose A State, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Include some patients in a second study to be developed
Supporting Information: SAP, ICF, CSR